CLINICAL TRIAL: NCT03667144
Title: Survival of Double Inlet Left Ventricle Patients Without Fontan Circulation: Intracardiac Anatomy and Hemodynamics, Functional Status and Quality of Life
Brief Title: Survival of Double Inlet Left Ventricle Patients Without Fontan Circulation
Acronym: DILV-S
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Groningen (Other)
Responsible Party: Principal Investigator, Sophie Meyer, Prof. dr. Tjark Ebels, University of Groningen
Other Study IDs: NL59516.042.17
Record Dates: First submitted 2018-08-15; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Double Inlet Left Ventricle
Keywords: Double inlet left ventricle without Fontan circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood samples for biomarker analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with univentricular hearts are currently palliated with the Fontan procedures. This results in an unphysiologic circulation with poor long-term survival. On the other hand there is a small, selected subgroup of patients with univentricular hearts of the double inlet left ventricle (DILV) type that survives up to old age without ever having undergone any Fontan procedures. Considering the relatively bleak data on long-term survival of DILV patients palliated with the Fontan procedure, it seems highly relevant to investigate and determine factors that allow a selection of unoperated patients to live to a comparatively high age without apparent major complaints. This might have an impact on how (and if, at all) certain univentricular patients are selected for operation in the future. For some, a different surgical procedure, or even therapeutic nihilism might be a more viable alternative.

The investigators hypothesise that favourable intracardiac streaming plays a role in making these patients viable: certain intracardiac anatomical characteristics allow for favourable flow patterns.

The primary objective of this study is to describe the intracardiac anatomy and hemodynamics of DILV patients without Fontan circulation using 4D MRI. Furthermore, the functional status and quality of life of these patients will be assessed.

DETAILED DESCRIPTION:
Rationale: Patients with univentricular hearts are currently palliated with a sequence of operations known as the Fontan procedure. This results in an un-physiologic circulation with poor long-term survival. On the other hand there is a small, selected subgroup of patients with univentricular hearts of the double inlet left ventricle (DILV) type that survives up to old age without ever having undergone any Fontan procedure. Considering the relatively bleak data on long-term survival of DILV patients palliated with the Fontan procedure, it is highly relevant to investigate and determine factors that allow for a selection of unoperated patients to live to a comparatively high age without apparent major complaints. This might have an impact on how (and if, at all) certain univentricular patients will be selected for operation in the future. For some, a different surgical procedure, or even therapeutic nihilism might be a more viable alternative. The investigators hypothesize that favourable intracardiac streaming plays a role in making the unpalliated patients viable: certain intracardiac anatomical characteristics allow for favourable flow patterns, resulting in higher systemic oxygen saturations than expected by mixing pulmonary and systemic venous returns.

Objective: The primary objective of this study is to describe the intracardiac anatomy and hemodynamics of DILV patients without Fontan circulation using 4D MRI. Furthermore, the functional status and quality of life of these patients will be assessed and compared to a matched cohort of Fontan patients.

Study design: This will be an observational, cross-sectional study. The investigators aim to include all DILV patients without Fontan circulation known at the congenital heart disease referral centers in the Netherlands and Flanders. The Dutch patients will undergo one 4D MRI, a physical examination, cardiopulmonary exercise testing and have a blood sample taken at the University Medical Center Utrecht. The patients from the Flemish referral centers will undergo the same protocol at the University Medical Center Leuven. Furthermore, patients over the age of 18 will be asked to fill out a quality of life questionnaire.

Study population: Included will be patients over the age of 12 with the diagnosis double inlet left ventricle, which have not undergone the Fontan trajectory. For the 4D MRI, patients with an MRI non-compatible pacemaker in situ will be excluded.

Main study parameters/endpoints: This is primarily an explorative study aiming to describe the anatomy of unpalliated DILV hearts of patients without Fontan palliation. With 4D MRI, the hearts will be grouped according to the angular relationship of the two lines connecting the atrioventricular and the ventriculo-arterial valves. This angle can be divided into three categories: 1) parallel (i.e. 0°), 2) perpendicular (i.e. 90°) or 3) an in-between variant. Accordingly, flow patterns, ranging from linear to turbulent will be measured and correlated to the anatomical variants.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden and risks associated with participation in this study are minimal. Patients need to visit the site of investigation only once, and the tests done at the visit (i.e. 4D MR imaging, exercise and pulmonary function testing and blood sample) are part of standard medical care and as such pose negligible risk on the patients. The quality of life survey is not part of standard medical care and might be confrontational on a psychological level. It is, however, a widely used and scientifically approved survey, which aims to keep this burden very low. Due to the extremely low prevalence of the condition to be studied, it is of great importance to include every single patient, including children under the age of 18. Excluding children from this study would further decrease the sample size to a significantly smaller number, making it difficult to draw conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis double inlet left ventricle, established by echocardiograph or MRI
* Not undergone Fontan trajectory in the past
* Be of the age of 12 or older
* Written informed consent

Exclusion Criteria:

• previous (partial) cavopulmonary connection

The following subjects will be excluded from the MRI part of the study, but will still be asked to participate in all the other parts:

• MRI non-compatible pacemaker in situ

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Included will be patients over the age of 12 with the diagnosis double inlet left ventricle, which have not undergone the Fontan trajectory. For the 4D MRI, patients with an MRI non-compatible pacemaker in situ will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-12-03 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Angle between atrioventricular and ventriculoarterial valves | 1 day
  This is primarily an explorative study aiming to describe the anatomy of unpalliated DILV hearts. With 4D MRI, the hearts will be grouped according to the angular relationship of the atrioventricular to the ventriculo-arterial valves. This angle can be divided into three categories: 1) parallel (i.e. 0°), 2) perpendicular (i.e. 90°) or 3) an in-between variant. Accordingly, flow patterns, ranging from linear to turbulent will be measured and correlated to the anatomical variants.

SECONDARY OUTCOMES:
New York Heart Association Functional Classification | 1 day
  NYHA functional class I to IV
Peak VO2 | 1 day
  peak oxygen uptake (VO2index) during exercise as well as peak VO2 as percentage of predicted (VO2 pred)
Peripheral oxygen saturation | 1 day
  Oxygen saturation at rest, measured with oximetry
Scores for Quality of life Adults | 1 day
  Quality of life survey overall scores, and scores in the subcategories measured with the Short Form (SF)36 (For patients 18 and older). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health
Scores for Quality of life | 1 day
  Quality of life survey overall scores, and scores in the subcategories measured with PedsQL (for patients younger than 18). The 23-item PedsQL Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. The 4 Multidimensional Scales are: Physical Functioning (8 items) Emotional Functioning (5 items), Social Functioning (5 items), School Functioning (5 items) The summary scores are: Total Scale Score (23 items), Physical Health Summary Score (8 items), Psychosocial Health Summary Score (15 items)
Hematocrit | 1 day
  from venous blood
Haemoglobin | 1 day
  from venous blood
Creatinin | 1 day
  from venous blood
eGFR | 1 day
  from venous blood
high sensitive Troponin T | 1 day
  from venous blood
NT-proBNP | 1 day
  from venous blood
LDH | 1 day
  from venous blood
ASAT | 1 day
  from venous blood
ALAT | 1 day
  from venous blood
Alkaline phosphatase | 1 day
  from venous blood
Gamma-GT | 1 day
  from venous blood
Galectin 3 | 1 day
  from venous blood
Bilirubin | 1 day
  from venous blood

OTHER OUTCOMES:
Demographics | 1 day
  sex, age, weight, height
Highest Level of Education | 1 day
  Highest level of education as well as their current Profession and their current work Status will be asked of all participants on the Basis of a questionnaire
Current Medication use | 1 day
  Participants will be asked to provide the names and the dosage of all medications they are currently using .

CONTACTS AND LOCATIONS:
Overall Officials: Tjark Ebels, MD PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frescura C, Thiene G. The new concept of univentricular heart. Front Pediatr. 2014 Jul 7;2:62. doi: 10.3389/fped.2014.00062. eCollection 2014. PMID 25072035
- [Background] Cook AC, Anderson RH. The anatomy of hearts with double inlet ventricle. Cardiol Young. 2006 Feb;16 Suppl 1:22-6. doi: 10.1017/S1047951105002283. No abstract available. PMID 16401359
- [Background] Franklin RC, Spiegelhalter DJ, Anderson RH, Macartney FJ, Rossi Filho RI, Douglas JM, Rigby ML, Deanfield JE. Double-inlet ventricle presenting in infancy. I. Survival without definitive repair. J Thorac Cardiovasc Surg. 1991 May;101(5):767-76. PMID 2023434
- [Background] Gersony WM. Fontan operation after 3 decades: what we have learned. Circulation. 2008 Jan 1;117(1):13-5. doi: 10.1161/CIRCULATIONAHA.107.748566. No abstract available. PMID 18172049
- [Background] Poterucha JT, Anavekar NS, Egbe AC, Julsrud PR, Connolly HM, Ammash NM, Warnes CA. Survival and outcomes of patients with unoperated single ventricle. Heart. 2016 Feb;102(3):216-22. doi: 10.1136/heartjnl-2015-308440. Epub 2015 Dec 23. PMID 26701967
- [Background] Macartney FJ, Partridge JB, Scott O, Deverall PB. Common or single ventricle. An angiocardiographic and hemodynamic study of 42 patients. Circulation. 1976 Mar;53(3):543-54. doi: 10.1161/01.cir.53.3.543. PMID 1248087
- [Background] Wolff D, van Melle JP, Bartelds B, Ridderbos FS, Eshuis G, van Stratum EBHJ, Recinos SJ, Willemse BWM, Hillege H, Willems TP, Ebels T, Berger RMF. Fontan Circulation over Time. Am J Cardiol. 2017 Aug 1;120(3):461-466. doi: 10.1016/j.amjcard.2017.05.005. Epub 2017 May 11. PMID 28624095
- [Background] Wolff D, van de Wiel HBM, de Muinck Keizer ME, van Melle JP, Pieper PG, Berger RMF, Ebels T, Weijmar Schultz WCM. Quality of life and sexual well-being in patients with a Fontan circulation: An explorative pilot study with a mixed method design. Congenit Heart Dis. 2018 Mar;13(2):319-326. doi: 10.1111/chd.12576. Epub 2018 Mar 12. PMID 29532606